CLINICAL TRIAL: NCT05720208
Title: Spinal Cord Innovation in Pediatrics (SCiP) to Treat SensoriMotor Function in Children Cerebral Palsy: Protocol for a Randomized Controlled Trial
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: SpineX Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: SPNX-02
Record Dates: First submitted 2023-01-31; First posted 2023-02-09 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-01

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapeutic Arm (Experimental)
  Interventions: Device: SCiP
- Sham Arm (Sham Comparator)
  Interventions: Device: SCiP

INTERVENTIONS:
Device: SCiP — Noninvasive Spinal Cord Neuromodulator

SUMMARY:
Cerebral palsy affects up to 4 children in 1000 live births, making it the most common motor disorder in children. It impairs the child's ability to move voluntarily and maintain balance and posture, and resultsing in a wide range of other functional disorders during early development that persist and frequently worsen with age including spasticity and often multiple abnormal sensationsensory modalities. Current standard of care treatments focus on symptom management and do not mitigate the progression of many of these underlying neurological impairments. The goal of this trial is to conduct a prospective multicenter, double-blinded, sham-controlled, crossover, randomized control trial to demonstrate the safety and efficacy of noninvasive spinal cord stimulation (using SCiPTM device, SpineX Inc.) in conjunction with activity-based neurorehabilitation therapy (ABNT) to improve voluntary sensorimotor function in children with cerebral palsy. 44 children participants (aged 2-18 years) diagnosed with CP classified as Gross Motor Function Classification Scale Levels I-V will be recruited and divided equally into two groups (G1 and G2). Both groups will receive identical ABNT 2 days/wk. G1 will initially receive sham stimulation, whereas G2 will receive therapeutic SCiPTM therapy for 8 weeks. After 8 weeks, G1 will cross over and receive therapeutic SCiPTM therapy for 8 weeks, whereas G2 will continue to receive SCiPTM therapy for another 8 weeks, for a total of 16 weeks. Primary and secondary outcome measures will include Gross Motor Function Measure-88 and Modified Ashworth Scale respectively.

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥ 2 and ≤ 18 years old at the time of enrollment/consent.
* Subject has a diagnosis of CP classified as Gross Motor Classification Scale Levels I-V.
* Minimum score of 12 and Maximum score of 85 on the GMFM-88 total score scale.
* Subject must have spastic CP hemiplegia or diplegia, quadriplegia.
* Subject's medical condition is stable as determined by the investigator.
* Subject has adequate social support network to be able to participate in training and assessment sessions for the duration of the study, at the discretion of the Investigator.
* Subject is capable of performing simple cued motor tasks and can follow 2-3 step commands.
* Subject can communicate an accurate yes or no answer to questions according to parents.

Exclusion Criteria:

* Subject has a concurrent neurological disease affecting the central nervous system.
* Subject has implanted stimulator (e.g., epidural stimulator, vagus nerve stimulator, pacemaker, cochlear implant, etc.) or drug delivery device (e.g., baclofen pump)
* Subject is dependent on an electro-magnetic medical implant (e.g., cardiac pacemaker or implanted drug pump), ventilation support, or another external device.
* Subject has received botulinum toxin injection within 12 months preceding enrollment.
* Subject is unable to participate in ABNT without orthosis.
* Subject has limited life expectancy or co-morbid conditions, social/psychological problems, or cognitive impairments that, in the opinion of the investigator, will preclude them from participation and completion of study procedures or requirements.
* Subject has a medical condition or complications related to the use of certain medications that may affect validity of the study as determined by the investigator.
* Subject has a medical condition not listed above that may put the subject at risk as determined by the investigator.
* Subject is participating in or plans to participate in another research study that may interfere with study endpoints.
* Subject is known or suspected to be non-compliant; and/or subject is unable or unwilling to comply with study requirements.
* Subject has cardiovascular or musculoskeletal disease or injury that would prevent full participation in physical therapy intervention
* Subject has a history of uncontrolled seizures.
* Subject has unhealed fracture or other musculoskeletal impairment that might interfere with upper or lower extremity rehabilitation or testing activities.
* Subject has a history of orthopedic surgery in upper or lower extremities or neurosurgery that may be a confounding factor for interpretation of the results (such as tendon transfer, tendon or muscle lengthening for spasticity management, injection therapies to lower extremity muscles, percutaneous lengthening, spinal fusion etc.) in last 12 months.
* Subject has a true leg length discrepancy greater than 2 cm.
* Subject has established osteoporosis and taking medication for osteoporosis treatment.
* Subject has undergone selective dorsal rhizotomy surgery.
* Subject has hip or shoulder migration percentage > 30% on anteroposterior radiographic imaging.
* Subject has less than 20 degrees in hip Range of Motion (ROM) in hip abduction.
* Subject has unexplained presence of persistent complaints of pain of any kind.
* Subject has fixed upper or lower extremity contractures of 20 degrees or more.
* Subject has a fixed spinal scoliosis greater than 20 degrees.
* Subject has severe cortico-visual impairment.
* Subject has other ongoing, or who has discontinued less than 14 days prior to consent, physical and occupational therapies including but not limited to robotic therapy, gait training, aqua therapy, hippo therapy, intensive therapies, whole body vibration (WBV), stimulation therapies (e.g., E-Stimulation, Functional Electrical Stimulation (FES), Neuromuscular Electrical Stimulation (NMES)).

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
GMFM88 | 8 weeks

SECONDARY OUTCOMES:
Modified Ashworth Scale | 8 weeks

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Girshin K, Sachdeva R, Cohn R, Gad P, Krassioukov AV, Edgerton VR. sPinal cOrd neUromodulatioN to treat Cerebral palsy in pEdiatrics: POUNCE Multisite Randomized Clinical Trial. Front Neurosci. 2023 Jul 26;17:1221809. doi: 10.3389/fnins.2023.1221809. eCollection 2023. PMID 37564370